CLINICAL TRIAL: NCT04326816
Title: Restorative Treatment of Severe Tooth Wear; Direct vs Indirect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/203
Record Dates: First submitted 2020-03-18; First posted 2020-03-30 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Tooth Wear; Dental Restoration Failure; Dental Restoration Wear
MeSH Terms: conditions — Tooth Wear | interventions — Clearfil AP-X

STUDY DESIGN:
Intervention Model Description: After written informed consent, patients fulfilling the inclusion criteria were assigned to an experimental group using block randomization with a block size of eight and the trial design had an intended allocation ratio of 1:1. Patients were allocated randomly to one of the two restorative treatment protocols: (1) Direct Composite restorations (DCR): using direct composite restorations on all teeth or (2) Indirect Composite Restorations (ICR): using ICR on all first molars and palatal veneer restorations on maxillary anterior teeth and DCR on remaining teeth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Composite Restorations (DCR) (Active Comparator): All teeth were reconstructed with directly applied composite restorations. No preparation of teeth was performed except in cases of sharp occlusal edges.
  Rubberdam or cotton rolls and suction devices were used for moisture control. For bonding, a 3-step etch-and-rinse adhesive was applied according to manufacturer's instructions, using 37% phosphoric acid (DMG, Hamburg, Germany), Clearfil SA Primer, and Clearfil Photobond (Kuraray, Osaka, Japan). A micro-hybrid composite (Clearfil AP-X, Kuraray) was used for posterior restorations and palatal veneer restorations. Restorations were placed according to the DSO-technique (Direct Shaping by Occlusion). In front teeth, both a palatal and buccal veneer restoration was placed.
  Experimental restorations were all restorations on first molars and all palatal veneer restorations on maxillary anterior teeth.
  Interventions: Procedure: Rehabilitation of severely worn dentitions using minimally invasive composite restorations (Estenia C&B or Clearfil AP-X, Kuraray, Osaka, Japan)
- Indirect Composite Restorations (ICR) (Experimental): Indirect 'tabletop' restorations were placed on all first molars (n=4) and palatal veneers ('backings') (n=6) on maxillary anterior teeth. Remaining teeth received directly applied restorations. Preparation of teeth for indirect restorations was limited to removal of sharp edges.
  All indirect restorations were laboratory manufactured using a micro-hybrid composite (Clearfil Estenia C&B, Kuraray, Osaka, Japan). Adhesive surfaces of the restorations were air-abraded with aluminum-oxide powder (<50 µm). Rubberdam or cotton rolls were used for moisture control during cementation. Seating of indirect restorations was checked intraorally, followed by cleaning of its adhesive surface with phosphoric acid 37% and application of silane (Clearfil Ceramic Primer, Kuraray, Osaka Japan).The adhesive surface of the abutment tooth was etched with phosphoric acid and ED-primer II (Kuraray) was applied. Finally, restorations were cemented, using Panavia F (Kuraray).
  Interventions: Procedure: Rehabilitation of severely worn dentitions using minimally invasive composite restorations (Estenia C&B or Clearfil AP-X, Kuraray, Osaka, Japan)

INTERVENTIONS:
Procedure: Rehabilitation of severely worn dentitions using minimally invasive composite restorations (Estenia C&B or Clearfil AP-X, Kuraray, Osaka, Japan)

SUMMARY:
This study compares the survival rates of both direct and indirect resin-based composite restorations in the treatment of severe tooth wear.

DETAILED DESCRIPTION:
Tooth wear can lead to pain, discomfort and unsatisfying dental attractiveness and when severe, it can compromise the dentition's prognosis. Restorative therapies for treatment of severe tooth wear should be preferably minimally invasive and adhesive.

This study compares two different treatment techniques for severe tooth wear. The first technique is regarded as the 'standard' technique. This is a full rehabilitation using only direct composite restorations (AP-X, Kuraray, Japan).

The second technique comprises a full rehabilitation using both direct and indirect resin composite restorations (Estenia C&B, Kuraray, Japan). 10 indirect restorations are placed on specific elements i.e. first molars and palatal sides of all maxillary anterior teeth. Other elements are restored conform the direct protocol.

An important benefit for the patients is the rehabilitation of their worn dentitions. Functionality (teeth are less sensitive, improved chewing ability, better occlusal stability, etc) and aesthetics will be improved immediately after finishing the treatment.

Indirect techniques have the advantage of a superior control over form of restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients age of at least 18 years old.
* Generalized moderate to severe tooth wear (Tooth Wear Index (TWI) ≥ 2) with a patient demand for treatment (Smith 1984)
* Full dental arches, but one diastema due to one missing tooth in the posterior area was allowed.
* An estimated need for increase of vertical dimension of occlusion (VDO) of ≥3mm at the location of the first molars.

Exclusion Criteria:

* Limited mouth opening (<3.5cm).
* (History of) Temporomandibular dysfunction, periodontitis, deep caries lesions or multiple endodontic problems.
* Local or systemic conditions that would contra-indicate dental procedures.

Patients with specific individual risk factors, such as parafunctional habits of grinding/clenching or patients with GORD (Gastro Oesophageal Reflex Disease), were not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Failure level 1 | Failures 3 years after placement
  Number of replaced direct and indirect restorations in the treatment. The higher the number the worse the outcome.
Failure level 2 | Failures 3 years after placement
  Number of repaired direct and indirect restorations in the treatment. The higher the number the worse the outcome.
Failure level 3 | Failures 3 years after placement
  Number of refurbished direct and indirect restorations in the treatment due to material chippings. The higher the number the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bas Loomans, PhD, DDS, Study Director — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No